CLINICAL TRIAL: NCT00419068
Title: Trial of Adjunctive Vitamin D in Tuberculosis Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: British Lung Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-003562-42; EudraCT no: 2005-003562-42; REC ref: 06/Q0605/83
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol
Drug: Migliol Placebo Oil

SUMMARY:
The purpose of this study is to determine whether vitamin D enhances response to standard antibiotic treatment for pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Suspected smear positive pulmonary tuberculosis.
* Age 18 years or older.
* Written informed consent to participate.

Exclusion Criteria:

* Known intolerance of vitamin D or first-line anti-tuberculous therapy.
* Taking antituberculous therapy for more than six days in the six months preceding enrolment.
* Taking the following medication in the month preceding enrolment: oral corticosteroid therapy, immunosuppressant therapy or cytotoxic therapy.
* Taking the following medication at enrolment: benzothiadiazine derivatives, cardiac glycosides or antituberculous therapy other than rifampicin, isoniazid, pyrazinamide and ethambutol.
* Diagnosis of any of the following: sarcoidosis, hyperparathyroidism, nephrolithiasis, pulmonary silicosis, HIV infection, liver failure, renal failure or malignancy
* Infection with rifampicin-resistant organism (as demonstrated by rapid molecular testing)
* Biochemical disturbance at enrolment: serum corrected calcium >2.66 mmol/l, serum AST >120 IU/l, total serum bilirubin > 40 micromol/l or serum creatinine > 250 micromol/l
* Breastfeeding or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Time to sputum culture conversion

SECONDARY OUTCOMES:
Rate of bacillary kill
2-month culture conversion rate
Time to sputum smear conversion
Weight change
Radiographic response

CONTACTS AND LOCATIONS:
Overall Officials: Adrian R Martineau, MRCP, Principal Investigator — Queen Mary University of London; Christopher J Griffiths, FRCP FRCGP D Phil, Principal Investigator — Queen Mary University of London
Locations (4):
- United Kingdom (4):
  - Whipps Cross University Hospital NHS Trust, London
  - Newham University Hospital NHS Trust, London
  - London Chest Hospital, London
  - Homerton University Hospital NHS Foundation Trust, London

REFERENCES:
- [Derived] Martineau AR, Timms PM, Bothamley GH, Hanifa Y, Islam K, Claxton AP, Packe GE, Moore-Gillon JC, Darmalingam M, Davidson RN, Milburn HJ, Baker LV, Barker RD, Woodward NJ, Venton TR, Barnes KE, Mullett CJ, Coussens AK, Rutterford CM, Mein CA, Davies GR, Wilkinson RJ, Nikolayevskyy V, Drobniewski FA, Eldridge SM, Griffiths CJ. High-dose vitamin D(3) during intensive-phase antimicrobial treatment of pulmonary tuberculosis: a double-blind randomised controlled trial. Lancet. 2011 Jan 15;377(9761):242-50. doi: 10.1016/S0140-6736(10)61889-2. Epub 2011 Jan 5. PMID 21215445